CLINICAL TRIAL: NCT04249648
Title: BuRden of Hyperkalaemia and EValuatIon of ChangEs to Therapy with Renin-angiotensin-aldosterone System Inhibitors Following Episodes of Elevated Potassium
Brief Title: Hyperkalaemia and Its Impact on Therapy with RAASi
Acronym: REVIEW
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Collaborators: Vifor Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: PHT/2020/11
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Hyperkalaemia; Heart Failure with Reduced Ejection Fraction; Left Ventricular Systolic Dysfunction
Keywords: Hyperkalaemia; Heart failure with reduced ejection fraction; Renin-angiotensin-aldosterone system inhibitors; Left Ventricular Systolic Dysfunction; Decision making process; Hyperkalaemia due to RAASi
MeSH Terms: conditions — Hyperkalemia; Ventricular Dysfunction, Left

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Patients with new diagnosis of heart failure with reduced ejection fraction: Patients with new diagnosis of heart failure with reduced ejection fraction who will be started on renin-angiotensin-aldosterone system inhibitors or in whom there is a plan to increase renin-angiotensin-aldosterone system inhibitors (if already taking prior to diagnosis of heart failure).
- Patients with hyperkalaemia: Hospitalised patients and patients attending emergency department who have at least 1 blood test with a potassium level of ≥5.5 mmol/l.
- Healthcare professionals managing patients with hyperkalaemia: Healthcare professionals (doctors, pharmacists, non-medical prescribers) who manage patients with hyperkalaemia and/or heart failure and hyperkalaemia.

SUMMARY:
Renin-angiotensin-aldosterone system inhibitors (RAASi) have transformed prognosis of patients with heart failure with reduced ejection fraction, diabetic nephropathy and chronic kidney disease. However, in everyday clinical practice patients often receive suboptimal doses of RAASi. The development of hyperkalaemia is one of the reasons for dose reduction or complete withdrawal of RAASi and this in turn is likely to have an adverse impact on patient outcomes. Yet it remains unknown precisely how often hyperkalaemia leads to changes to RAASi doses, if it is the sole reason, or whether this occurs in combination with other clinical situations such as worsened renal function and hypotension. It is also unclear what influences the decision-making process of healthcare professionals in managing patients with hyperkalaemia who take RAASi and if this is influenced by specialty, experience or indications for RAASi.

In order to improve our understanding of the problem we are taking forward a research study (made up of 3 complimentary studies). These data are needed to help achieve our ultimate goal of improving the care of patients with prognostic indication for RAASi.

DETAILED DESCRIPTION:
The study aims to answer the following research questions:

1. What is the incidence of hyperkalaemia following RAASi therapy initiation and uptitration in patients with a new diagnosis of HFrEF including those with a new diagnosis of post myocardial infarction (MI) left ventricular systolic dysfunction?
2. How does it impact on RAASi prescription?
3. How does hyperkalaemia impact on RAASi therapy according to the clinical indication for the drug(s) in an adult population of patients who are hospitalised or attending the emergency department (and not receiving dialysis) with hyperkalaemia and receiving RAASi?
4. At what level of hyperkalaemia do healthcare professionals consider making changes to RAASi and does it vary according to the clinical indication for the drug(s)?

ELIGIBILITY:
For patients with heart failure

Inclusion criteria

1. Patients with newly diagnosed HFrEF (within 4 weeks of diagnosis, including those with post MI LVSD, identified as outpatients or during hospital admission, typically for decompensated heart failure or post myocardial infarction) who are initiated on RAASi or have a clinical indication for uptitration of current RAASi (in patients already receiving RAASi for other indications).
2. Able to provide informed consent.
3. Age 18 and above.

Exclusion criteria: 1. Patients receiving dialysis.

For patients with hyperkalaemia

Inclusion criteria

1. Patients in ED or inpatients who already receive RAASi and who have at least 1 blood test with a potassium level of ≥5.5 mmol/l.
2. Able to provide informed consent.
3. Age 18 and above.

Exclusion criteria: 1. Patients receiving dialysis.

For healthcare professionals:

Inclusion criteria

1. Doctors, pharmacists, non-medical prescribers working at primary and secondary care.
2. Able to provide informed consent.
3. Age 18 and above.

Exclusion criteria: 1. None

As this is an observational study, patients in other research studies or receiving any specific treatments for hyperkalaemia (other than chronic dialysis) will not be excluded. After consent, patients will also be permitted to participate in other research studies should they so wish. Patients with covid-19 can also be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed heart failure with reduced ejection fraction (within 4 weeks of diagnosis, including those with post myocardial infarction left-ventricular systolic dysfunction)
  Patients in ED or inpatients who already receive RAASi and who have at least 1 blood test with a potassium level of ≥5.5 mmol/l and not receiving dialysis prior to the episode of hyperkalaemia.
  Healthcare professionals managing patients with hyperkalaemia and/or heart failure
Sampling Method: Non-Probability Sample
Enrollment: 651 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Incidence of hyperkalaemia in patients with new diagnosis of HFrEF | 12 months
  Incidence of hyperkalaemia in patients with new heart failure with reduced ejection fraction started on renin-angiotensin-aldosterone receptor inhibitor(s)
Frequency of dose reduction/withdrawal for RAASi after hyperkalaemia in patients with HFrEF | 12 months
  Proportion of patients with new HFrEF started on RAASi who experienced RAASi dose reduction/withdrawal/prevention of dose uptitration due to hyperkalaemia.
Proportion of patients with hyperkalaemia (hospitalised or attending ED) who experienced changes to RAASi after episodes of hyperkalaemia | 12 months
  3. Proportion of hospitalised patients/ED attenders with documented hyperkalaemia, receiving RAASi for prognostic benefit who experience RAASi dose reduction/withdrawal, assessed at discharge

SECONDARY OUTCOMES:
Incidence of repeated episodes of hyperkalaemia | 12 months
  Incidence of repeated episodes of hyperkalaemia after initial episode.
RAASi discontinuation due to other causes rather than hyperkalaemia | 12 months
  Proportion of patients discontinuing RAASi due to other causes than hyperkalaemia (hypotension, worsening renal function, other).
Mortality | 12 months
  Number and causes (all cause, cardiovascular or HF) of mortality at 12 months.
Hospitalisations | 12 months
  Number and causes (all cause, cardiovascular or HF) of hospitalisation at 12 months.
Hyperkalaemia level at which healthcare professionals make changes to RAASi | 12 months
  Level of hyperkalaemia at which healthcare professionals reduce/stop RAASi in patients with and without clear prognostic indications for RAASi.
Description of healthcare professionals making changes to RAASi after episodes of hyperkalaemia | 12 months
  Proportion of different grades and specialties of healthcare professionals reducing dose/stopping RAASi in hyperkalaemic patients.
Awareness of RAASi benefits and target doses for patients with HFrEF | 12 months
  Proportion of different grades and specialties of healthcare professionals who are aware of RAASi target doses and benefits in HFrEF.

CONTACTS AND LOCATIONS:
Overall Officials: Paul R Kalra, Professor, Principal Investigator — Queen Alexandra Hospital, Portsmouth, UK
Locations (1):
- Portsmouth Hospitals University NHS Trust, Portsmouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan to share IDP